CLINICAL TRIAL: NCT00706459
Title: Advanced MR Imaging in Patients With Painful, Degenerative Disc Disease: A Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Due to funding issue, study has been terminated.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: SpineMRI
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Disc specimens are taken out during back surgery and will be studied using techniques for tissue analysis to explain the properties and characteristics of disc tissue from patients with back pain.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Patients with lumbar back pain scheduled for back surgery.
  Interventions: Device: Magnetic Resonance Imaging
- 2: Patients with degenerative disease without classic discogenic back pain
  Interventions: Device: Magnetic Resonance Imaging
- 3: Normal control without back pain.
  Interventions: Device: Magnetic Resonance Imaging
- 4: Post Surgical discectomy patients
  Interventions: Device: Magnetic Resonance Imaging
- 5: disc specimens
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — All study subjects will have a 3T MRI examination. The MRI exam will take approximately 90 minutes to complete and will involve the scanning o the spine.

SUMMARY:
In this study, we will use advanced and newly available MR imaging techniques at 3 Tesla (including in situ axial loading and quantitative T1rho, T2, and diffusion measurements) to assess the intervertebral discs and adjacent vertebrae in patients with lumbar back pain scheduled for back surgery (n=20), patients with degenerative disease without classic discogenic back pain (n=10), patients who had discectomies for herniated discs (n=5), and age-matched volunteers without back pain (n=10). In all patients standard imaging procedures will also be performed, including radiographs, standard MRI at 1.5 Tesla and discography. All patients will have specimen of the intervertebral disc harvested at surgery and pathologic analysis and spectroscopy of these specimen will be performed. Post-surgical findings/outcome combined with discography will serve as a standard of reference for the identification of the painful disc(s). The diagnostic performance of the new techniques in assessing the painful disc will be evaluated. We will collect disc specimens from 50 patients undergoing back surgery but did not have pre-surgical MR imaging. These disc specimens will be analyzed in the same manner as the specimens collected from surgical patients who had pre-surgical MRI. This study will serve as a pilot study for a larger project focusing on advanced imaging of the painful intervertebral disc.

We hypothesis that advanced, dedicated MR examinations at 3T can identify painful degenerated discs in patients with chronic lumbar back pain.

ELIGIBILITY:
Inclusion Criteria for Patient with classic discogenic back pain:

* age range 25-60 years old
* Back and/or leg (back>leg) pain
* Degenerative disc disease in one or more adjacent vertebral levels between L3-S1
* Radiologic confirmation of degenerative disc disease:
* Segmental instability (3 mm translation or 5 degree angulation)
* Decreased disc height >2 mm
* Scarring, thickening of annulus fibrosis
* Vacuum phenomenon
* No significant foraminal stenosis and nerve root compression
* Failed observative treatment for at least 6 months
* Oswestry LB disability questionnaire score of at least 20/50 (40%) (interpreted as moderate to severe disability)
* Psychosocially and mentally normal
* Patients who are scheduled for back surgery

Inclusion criteria for patients with degenerative disc disease without the classic discogenic back pain:

* Age range 25-60 years old
* Patients with diagnosis of idiopathic scoliosis, spondylolysis, or spondylolisthesis

Inclusion criteria for normal controls:

* No symptoms
* Age range 25-60 years old

Inclusion Criteria for post-surgical discectomy patients:

* Patients who had successful disc surgery for lumbar herniated disc and no further back pain
* Patients who had unsuccessful disc surgery for lumbar herniated disc and still with residual back pain

Exclusion Criteria:

* prior back surgery (except as mentioned above)
* spine fractures
* Radiographic confirmation of facet joint disease or degeneration
* Radiographic confirmation of sacroiliac joint pathology
* Lytic spondylolisthesis of spinal stenosis
* Degenerative spondylolisthesis of > grade 1
* Metabolic bone disease
* Spine infection , osteomyelitis
* Rheumatoid arthritis or any other systemic or autoimmune disease
* Active malignancy
* MRI Contraindications (fragment in eye, aneurysms clips, ear implants, spinal nerve stimulators, pacemaker, claustrophobia, or pregnant women, etc.,)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Potential subjects are patients seen by surgeons in the UCSF ACC Orthopedic Clinic. If a patient meets all inclusion and exclusion criteria, the orthopedic surgeon will talk to the patient about the new dedicated examinations using 3 Tesla MRI that can identify painful degenerated discs. When patient is comfortable with participating and has made a decision to go ahead with the MRI, patient can let the orthopedic surgeon's assistant know about his/her decision, the assistant will make sure that patient still meets the inclusion and exclusion criteria and will call the coordinator at the Imaging Center to set up an MRI appointment.
  Flyers will be posted at different UCSF campuses to recruit for normal age-matched and young normal volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2005-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Majumdar, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States